CLINICAL TRIAL: NCT01537705
Title: A Clinical Outcomes Study to Measure Reduction in Pain and Numbness During Administration of an Amino Acid Formulation in Subjects Diagnosed With Peripheral Neuropathy
Acronym: Neuron012703
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Targeted Medical Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012703
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Diabetic Neuropathy; Chemotherapy Induced Neuropathy; HIV Neuropathy; Trauma Induced Neuropathy
Keywords: Medical food; Neuropathy; Diabetes; Neuropathic Pain
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neuron012703 (Experimental): Amino acid formulation for the dietary management of symptoms related to periphal neuropathy.
  Interventions: Drug: Neuron012703 (Medical Food)

INTERVENTIONS:
Drug: Neuron012703 (Medical Food) — 2 capsules twice daily for sixty days.

SUMMARY:
A clinical outcomes study measuring reduction in pain and numbness experienced in four types of peripheral neuropathy patients during 60 day administration of the an amino acid formulation.

DETAILED DESCRIPTION:
Peripheral neuropathy is a disorder of the peripheral nerves-the motor, sensory and autonomic nerves that connect the spinal cord to muscles, skin and internal organs. It usually affects the hands and feet, causing weakness, numbness, tingling and pain. Peripheral neuropathy's course is variable; it can come and go, slowly progressing over many years, or it can become severe and debilitating. Peripheral neuropathy is common and it is estimated that upwards of 20 million Americans suffer from this illness. It can occur at any age, but is more common among elderly patients. In l999, a survey found that 8-9% of Medicare recipients have peripheral neuropathy as their primary or secondary diagnosis and the annual cost to Medicare exceeds $3.5 billion. Approximately 30% of peripheral neuropathy cases are linked to diabetes. Other common causes of neuropathy include autoimmune disorders, tumors, hereditary conditions, nutritional imbalances, infections or toxins. Another 30% of peripheral neuropathies are termed "idiopathic" when the cause is unknown. Pain in particular is a complex process initiated by pain-inducing or noxious stimuli interacting with pain receptors (nociceptors) which triggers a series of action potentials that are transmitted by neurotransmitters from peripheral afferent neurons to the spinal cord and higher nerve centers in the brain.

The study intervention is classified as a medical food that must be used under the active or ongoing supervision of a physician. Medical foods are developed to address the different or altered physiologic requirements that may exist for individuals with distinctive nutritional needs arising from metabolic disorders, chronic diseases, injuries, premature birth associated with inflammation and other medical conditions, as well as from pharmaceutical therapies. All of the ingredients included in the study intervention are classified as generally recognized as safe (GRAS) by the United States Food and Drug Administration (FDA). To qualify for GRAS status, a substance that is added to a food, including a medical food, has to be supported by data demonstrating that it is safe when consumed in amounts from these foods, as they are typically ingested or prescribed.

The study intervention is a proprietary blend of amino acids and antioxidants designed to target the cellular processes involved in the management of peripheral neuropathy symptoms. All of the ingredients are supplied in small milligram quantities which allows for safe and flexible dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of peripheral neuropathy diagnosis from physician.
2. Subjects able to read and understand English.
3. Subjects willing to commit to all study visits for the duration of administration.
4. Male and non-pregnant/lactating females, ages 18 to 75.

Exclusion Criteria:

1. Subjects hospitalized within the last 30 days.
2. History of nerve surgery.
3. Currently taking other medical foods.
4. Existing serious medical condition (i.e. severe heart, liver or kidney disease).
5. Subjects with measured creatinine greater than 2.5, ALT or AST greater than three times normal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
VAS | 60 Days
  To measure reduction in pain related to various types of peripheral neuropathy during administration of study intervention using a Visual Analog Scale.

SECONDARY OUTCOMES:
NTSS-6 | 60 Days
  Neuropathy Total Symptom Score-6
Routine Blood Panel | 60 days
  CBC, Liver panel

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Halperin, DPM, Principal Investigator — Gabriel Halperin DPM Inc.
Locations (1):
- Gabriel Halperin DPM Inc, Los Angeles, California, United States